CLINICAL TRIAL: NCT05916508
Title: A One-Month Bleeding-Model Clinical Study
Brief Title: A Bleeding-Model Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020112
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis | interventions — Tin Fluorides; fluorophosphate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Positive Control (Active Comparator): 2 brushings per day (AM and PM)
  Interventions: Drug: 0.454% stannous fluoride
- Negative Control (Sham Comparator): 2 brushings per day (AM and PM)
  Interventions: Drug: 0.76% sodium monofluorophosphate
- Experimental Control (Experimental): Brush with Positive control in the morning and negative control in the evening
  Interventions: Drug: 0.454% stannous fluoride AM and 0.76% sodium monofluorophosphate PM

INTERVENTIONS:
Drug: 0.454% stannous fluoride — Brush two times daily
  Arms: Positive Control
Drug: 0.76% sodium monofluorophosphate — Brush two times daily
  Arms: Negative Control
Drug: 0.454% stannous fluoride AM and 0.76% sodium monofluorophosphate PM — Brush two times daily
  Arms: Experimental Control

SUMMARY:
The objective of the study is to evaluate the gingivitis control benefit of an established stannous fluoride containing toothpaste relative to a negative control dentifrice.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age;
* Provide written informed consent prior to participation and be given a signed copy of the informed consent form;
* Be in general good health as determined by the Investigator based on a review of the health history/update for participation in the trial;
* Have at least 20 gradable teeth;
* Have established gingivitis with ≥10 % bleeding sites;
* Agree to return for scheduled visits and follow the study procedures;
* Agree to refrain from use of any non-study oral hygiene products for the duration of the study;
* Agree to delay any elective dentistry, including dental prophylaxis, until the completion of the study.

Exclusion Criteria:

* Having taken medications (antibiotic, anti-inflammatory, or anti-coagulant) which could alter gingival bleeding within 4 weeks of the Baseline Visit;
* Having any oral conditions that could interfere with study compliance and/or examination procedures, such as widespread caries, soft or hard tissue tumor of the oral cavity, or advanced periodontal disease;
* Having known hypersensitivity to the test products;
* Having removable oral appliances;
* Having fixed facial or lingual orthodontic appliances;
* Self-reported pregnancy or lactation;
* Having any diseases or condition that might interfere with the safe participation in the study;
* Having an inability to undergo study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Löe-Silness Gingivitis Evaluation | Baseline
  Löe-Silness Gingivitis Evaluation is a validated assessment of gingival health looking at inflammation and bleeding based on a 4 point range 0 (normal gingiva) to 3 (severe inflammation).
Löe-Silness Gingivitis Evaluation | Week 4
  Löe-Silness Gingivitis Evaluation is a validated assessment of gingival health looking at inflammation and bleeding based on a 4 point range 0 (normal gingiva) to 3 (severe inflammation).

CONTACTS AND LOCATIONS:
Locations (1):
- Silverstone Research Group, Las Vegas, Nevada, United States

REFERENCES:
- [Derived] He T, Zou Y, Grender J, Amini P, Kaminski M, Biesbrock AR. Randomized Controlled Trials Assessing Exposure Frequency Effects of Stannous Fluoride on Gingivitis. JDR Clin Trans Res. 2025 Apr;10(2):124-134. doi: 10.1177/23800844241263031. Epub 2024 Aug 8. PMID 39118360